CLINICAL TRIAL: NCT05254509
Title: The Effects of Virtual Reality With Debriefing on Patients With Chronic Pain
Brief Title: Virtual Reality, Debriefing and Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Ajay Wasan, MD, Msc, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY21110066
Record Dates: First submitted 2022-02-23; First posted 2022-02-24 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Chronic Pain
Keywords: chronic pain; virtual reality; Occupational therapy; debriefing; self-efficacy; fear of movement
MeSH Terms: conditions — Chronic Pain; Kinesiophobia | interventions — Occupational Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Occupational Therapy (OT) (Active Comparator): Subjects in this treatment group will receive outpatient occupational therapy geared towards people with chronic pain conditions. After obtaining consent, an occupational therapist will meet with the participant to begin their occupational therapy sessions targeted for those who have chronic pain. Additionally, subjects will complete online surveys administered by the therapist before and after each therapy session. There is a total of six 1-hour visits during the 3-month study duration involving occupational therapy. They will also receive online surveys every two weeks and will be asked to complete them at home.
  Interventions: Other: Occupational Therapy
- Occupational Therapy + Virtual Reality (OT+VR) (Experimental): Subjects in this treatment group will receive outpatient occupational therapy intervention geared towards people with chronic pain conditions followed by active, immersive virtual reality sessions. Participants in this treatment group will have 10-30minutes of usual care while receiving 10-30 minutes of virtual reality (e.g. exercises, games, and activities in the virtual world) during each study visit. Subjects will complete online surveys before and after each virtual reality session, along with debriefing from a therapist after each VR session to review what happened and why. Debriefing will include questions to obtain thoughts and narrative information about the participant's experience, as well as overall take-aways from the session. The therapist and subject will also watch a video recording of the subject's VR experience as a method to provide them feedback on their performance. Subjects will receive online surveys every two weeks and will be asked to complete them at home.
  Interventions: Other: Occupational Therapy +Virtual Reality

INTERVENTIONS:
Other: Occupational Therapy — Occupational therapy helps individuals with chronic pain to participate in daily activities in an adaptive way. The subjects will be provided with customized plans and objectives to address their self-care, vocational, and leisure goals. This includes education, home exercises, stress management, home safety, energy conservation, and work simplification - all of which promote a safe return to daily activities.
  Other Names: OT
  Arms: Occupational Therapy (OT)
Other: Occupational Therapy +Virtual Reality — The occupational therapy +VR utilizes the regular therapy sessions along with providing a Virtual reality headset to relieve pain. After each VR session, there will be a debriefing from the therapist.
  Other Names: OT+VR
  Arms: Occupational Therapy + Virtual Reality (OT+VR)

SUMMARY:
This study will determine if occupational therapy or the combination of occupational therapy and virtual reality is the better treatment for chronic low back pain (CLBP)patients.

DETAILED DESCRIPTION:
Chronic musculoskeletal pain is defined as persistent or recurrent pain lasting more than 3 months. Chronic pain is a complex and disabling physiological and psychosocial disorder that does not provide an adaptive or protective purpose. In chronic pain, the precipitating event (e.g., fracture, sprain, trauma) is healed, and yet excessive pain remains. In Immersive Virtual Reality (IVR) people experience a three-dimensional, computer-generated environment via a computer headset. IVR has been used to treat acute pain, but there have been few focused studies on the effects of IVR on chronic pain. When people with chronic pain are in IVR, they become unaware of their body and tend to move normally. We would like to test to see if IVR has a lasting effect in this study. Thus, IVR has strong potential as an additional tool in an arsenal of treatments for chronic pain. This study will examine if IVR can reduce pain and other symptoms in people with chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 and older
* Referred for chronic pain occupational therapy services at the UPMC Centers for Rehab Services Centre Commons site.

Exclusion Criteria:

* Had a seizure, loss of awareness, or other symptom linked to an epileptic condition
* Had virtual reality intervention within the last 3 months
* Has sensory insensitivity such as hearing loss or low vision, as assessed by the PI
* Has contagious disorder on the face, such as pink eye, that could be transmitted via the VR headset or has open areas on the face that would come in contact with the headset
* Has a pacemaker or defibrillator
* Insufficient upper extremity coordination to operate IVR controls, as assessed by the PI
* Insufficient cognitive ability to answer questionnaires or learn to use the IVR, as assessed by the PI
* Have a diagnosis of ASD (Autism Spectrum Disorder) or unable to understand and/or respond in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-04-18 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-09-13 (Actual)

PRIMARY OUTCOMES:
Changes from Baseline in average rating of chronic pain at 3 months using Numeric Pain Rating Scale | Baseline vs 3 months
  Numeric Pain Rating questionnaire will assess how much a person hurts with a question ranked on a 11-point scale, from "0 = no pain" to "10 = worst pain imaginable." The minimum raw summed score is 0 and the maximum score is 10. Lower raw response scores suggest lower pain intensity and better outcomes.

SECONDARY OUTCOMES:
Change from Baseline self-efficacy using Pain Self Efficacy Questionnaire (PSEQ). | Baseline vs 3 months
  Change from Baseline Pain Self Efficacy at 3 months using Pain Self Efficacy Questionnaire (PSEQ). The questionnaire will assess how confident a person feels despite the pain with 10 questions ranked on a 7-point scale, from "0 = not at all confident" to "6 = Completely confident".
Change from Baseline fear of movement using the Tampa Scale of Kinesiophobia (TSK). | Baseline vs 3 months
  The Tampa Scale of Kinesiophobia (TSK) questionnaire will assess fear of movement with 17 questions ranked on a 1-4 scale, from "1 = Strongly disagree" to the "4 = Strongly agree." Lower scores suggest lower fear of movement.
Change from Baseline Pain Intensity at 3 months using PROMIS-29 | Baseline vs 3 months
  The PROMIS Numeric Rating Scale v2.0 questionnaire will assess how much a person hurts with a question ranked on a 11-point scale, from "0 = no pain" to "10 = worst imaginable pain." The minimum raw summed score is 0 and the maximum score is 10. Lower raw response scores suggest lower pain intensity and better outcomes.
Change from Baseline participation and scaling at 3 months using Goal Attainment Scale (GAS) | Baseline vs 3 months
  The Goal Attainment Scale will assess the response to participation based on a 5 point scale ranging from "+2 = MUCH more than expected" to "-2 = MUCH less than expected".HIgher scores suggest higher response to participation.

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Wasan, MD,MSc, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Centers for Rehab Services Centre Commons, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No